CLINICAL TRIAL: NCT04843930
Title: Improving Cognitive Health in COVID-19 Survivors Through Digital Therapeutics
Brief Title: Improving Cognitive Health in COVID-19 Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-11022977
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Dysfunction; Covid19
Keywords: Covid19; Cognitive Dysfunction; Attention Disturbances; Cognitive Change
MeSH Terms: conditions — Cognitive Dysfunction; COVID-19

STUDY DESIGN:
Intervention Model Description: This study is a randomized clinical trial designed to compare efficacy of the AKL-T01 intervention relative to a waitlist control in patients who were infected with COVID-19. Participants will be randomized to the AKL-T01 or a waitlist control. We will use a waitlist design; at the end of the intervention period, participants in the control group will have the option to receive the 6-week AKL-T01 intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care managers will be instructed not to reveal the group assignment to the member of the research team conducting assessments. Following the completion of recruitment, data analysts will be provided with the data for the arms simply labelled as "Group A" and "Group B" to avoid bias. These generic labels will be unmasked only after completion of all the planned statistical analyses described below. Participants in the waitlist control arm who begin the intervention at the end of the waitlist period will have different assessors for the initial 6-week control procedures and the subsequent 6-week intervention period so as to maintain the blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AKL-T01 Intervention (Experimental): Participants in the experimental group will complete 6 weeks of the AKL-T01 intervention. Participants enrolled in the intervention arm will play the game via an iPad application for 20-25 minutes daily for at least 5 days a week (but up to 7 days a week). Participants will also have weekly check-in visits via phone or a secure HIPAA compliant videoconferencing platform (Zoom) with a care manager, who will monitor mood symptoms and gameplay adherence.
  Interventions: Device: AKL-T01
- Waitlist Control (No Intervention): Participants in the Waitlist Control arm will not be engaging in any active control condition. Participants in the waitlist control arm will continue any ongoing self- or provider-based cognitive intervention (or no intervention) during the initial 6-week waitlist period. Participants will also have weekly check-in visits via phone or a secure HIPAA compliant videoconferencing platform (Zoom) with a care manager, who will monitor mood symptoms. The control arm will be offered the intervention at the end of 6 weeks waitlist period to ensure all participants ultimately have access to the intervention.

INTERVENTIONS:
Device: AKL-T01 — AKL-T01 will be administered as a 6-week intervention. It is an algorithmically delivered iPad-based video game designed to improve cognitive health by targeting attention and attentional control processes.
  Arms: AKL-T01 Intervention

SUMMARY:
The primary objective of this study is to investigate the efficacy of AKL-T01, a remotely-delivered digital cognitive intervention, relative to a waitlist control in improving cognitive functioning in COVID-19 survivors.

DETAILED DESCRIPTION:
Emerging evidence suggests a subgroup of survivors of COVID- 19 have residual difficulties with cognition and daily functioning. These deficits are pronounced in cognitive domains including attention, learning and executive skills, and may continue to impact quality of life after recovery from other COVID-19 symptoms. This study aims to investigate the efficacy of AKL-T01 (Akili Interactive), a remotely-delivered digital cognitive intervention, in targeting and improving cognition and functional outcomes in individuals recovering from COVID-19. The efficacy of the AKL-T01 intervention will be measured relative to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-89 years of age
* Documentation of a deficit in cognitive function (score > 1 standard deviation below normal range) compared to age-adjusted normative data) on at least one screening measure of attention and executive function (Oral Trail Making Test, Stroop Test, or FrSBe)
* Previous diagnosis of COVID-19 confirmed via SARS-CoV-2 polymerase chain reaction (PCR) test (or reported experience of COVID-19 symptoms with a documented positive antibody test or clinical diagnosis based on symptoms and accompanying physician's note) documented in the electronic medical record or in other existing medical records
* Access to and self-report of ability to connect wireless devices to a functional wireless network.
* Ability to follow written and verbal instructions (English) as assessed by the PI and/or coinvestigator.
* Able to comply with all testing and study requirements and willingness to participate in the full study duration

Exclusion Criteria:

* History of neurologic disorder prior to COVID-19 diagnosis, such as Parkinson's disease, multiple sclerosis, Alzheimer's disease, stroke, brain tumor, or dementia.
* History of severe mental illness (e.g., schizophrenia, psychosis, history of suicide attempt in the last year) or substance use disorder, recent history (in the past year) of symptoms of psychosis
* Participant is currently considered at risk for attempting suicide by the Investigator, has made a suicide attempt within the past year, or is currently demonstrating active suicidal ideation or self-injurious behavior.
* Motor condition (e.g., physical deformity of the hands/arms) that prevents game playing as reported by the participant or observed by the Investigator
* Recent history (within 6 months prior to screening/baseline) of substance use disorder
* History of seizures (excluding febrile seizures), a tic disorder, significant tics, a current diagnosis of Tourette's Disorder.
* Color blindness as determined by self-report
* Regular use of psychoactive drugs other than antidepressants or benzodiazepines, including stimulants that in the opinion of the Investigator may confound study data/assessments.
* Any other acute medical condition that may interfere with participation or interpretation of the results
* Previous exposure to AKL-T01.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gunning, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2021 (date of first enrollment: 7/13/2021) and December 2022 (date of final enrollment: 12/7/2022). Participants were recruited through facilities of the Manhattan Campuses of NewYork-Presbyterian Hospital (NYP)/Weill Cornell Medicine (WCM), as well as the NewYork-Presbyterian Westchester Behavioral Health Center. Participants were also recruited through community advertisement in the Greater New York City area.
Pre-assignment Details: Note that the final participant was consented and enrolled on 12/7/2022, but did not have their first study visit until 12/20/2022 due to scheduling constraints. The final 6-week primary endpoint for this participant was collected on 2/6/2023.
Groups:
- AKL-T01 Intervention: Participants in the intervention arm complete 6 weeks of the AKL-T01 intervention. Participants complete the intervention (an algorithmically delivered iPad-based video game designed to improve cognitive health by targeting attention and attentional control processes) for 20-25 minutes daily for at least 5 days a week (but up to 7 days a week). Participants also have weekly check-in visits with a care manager to complete assessments and monitor mood symptoms and gameplay adherence.
- Waitlist Control: Participants in the waitlist control arm will not be engaging in any active control condition. Participants will also have weekly check-in visits with a care manager to complete assessments and monitor mood symptoms. The control arm will be offered the intervention at the end of 6 weeks waitlist period to ensure all participants ultimately have access to the intervention.
- Control Arm Participants Who Started AKL-T01 Intervention: Participants who opted to start the intervention after the waitlist control period.
- Control Arm Participants Who Declined AKL-T01 Intervention: Participants who opted to not start the intervention after the waitlist control period.
Period: Randomization
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
Started | 55 | 55 | 0 | 0
Completed | 49 | 49 | 0 | 0
Not Completed | 6 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 0 | 0
Period: Baseline Assessment
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
Started | 49 | 49 | 0 | 0
Completed | 49 | 49 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Week 6 Assessment
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
Started | 49 | 49 | 0 | 0
Completed | 44 | 48 | 0 | 0
Not Completed | 5 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Period: Week 10 Follow-Up
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
Started | 44 | 0 | 0 | 2
Completed | 44 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2
Period: Week 16 Follow-Up
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
Started | 0 | 0 | 46 | 0
Completed | 0 | 0 | 44 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis includes the sample who initiated the trial and were included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | AKL-T01 Intervention | Waitlist Control | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (17.2) | 46.8 (16.7) | 48.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 5 | 8
  Black | 10 | 12 | 22
  Hispanic/Latinx | 6 | 4 | 10
  White | 25 | 23 | 48
  More Than One Race | 2 | 4 | 6
  Other / Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98
Education [Mean (Standard Deviation); unit: years] | 16.9 (2.8) | 16.7 (2.2) | 16.8 (2.5)
COVID Treatment Category [Count of Participants; unit: Participants]
  Outpatient | 16 | 12 | 28
  ER Admission | 2 | 4 | 6
  Inpatient | 1 | 2 | 3
  ICU | 3 | 5 | 8
  No Treatment | 26 | 21 | 47
  Other | 1 | 5 | 6
Oral Trails A [Mean (Standard Deviation); unit: seconds] — Assessment of executive function / sequential set shifting. Participants are instructed to count verbally from 1 to 25; the time to complete the count is recorded in seconds. Longer times indicate more executive dysfunction.
  seconds | 8.9 (2.6) | 8.3 (2.4) | 8.6 (2.5)
Oral Trails B [Mean (Standard Deviation); unit: seconds] — Assessment of executive function / sequential set shifting. Participants are instructed to count verbally from 1 to 13, alternating a number and a letter (e.g., 1-A-2-B-3-C, etc.); the time to complete the count is recorded in seconds. Longer times indicate more executive dysfunction.
  seconds | 32.0 (15.3) | 32.6 (16.5) | 32.3 (15.8)
Stroop Color-Word t-score [Mean (Standard Deviation); unit: t-score] — Stroop Task interference for incongruent color/word stimuli. Participants read color-word stimuli aloud for 45 seconds, score represents number of words read. Reported t-scores are corrected for age and education. Greater scores indicate less executive dysfunction. A t-score of 50 represents the population mean (with a standard deviation of 10). A t-score of 40 reflects performance one standard deviation below age- and education-adjusted norms (16th percentile). Participants that performed > or equal to one standard deviation below adjusted means were considered for inclusion in the trial.
  t-score | 39.6 (19.3) | 41.8 (19.5) | 40.7 (19.4)
FrSBe Total Score (before COVID) [Mean (Standard Deviation); unit: score on a scale] — Frontal Systems Behavior Scale, a self-report measure of apathy, disinhibition, and executive dysfunction. Scored on a scale from 46-230; higher score indicate more dysfunction.
  score on a scale | 79.5 (17.7) | 80.4 (16.4) | 79.9 (17.0)
FrSBe Total Score (after COVID) [Mean (Standard Deviation); unit: score on a scale] — Frontal Systems Behavior Scale, a self-report measure of apathy, disinhibition, and executive dysfunction. Scored on a scale from 46-230; higher score indicate more dysfunction.
  score on a scale | 111.0 (23.8) | 109.0 (20.8) | 110.0 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function, as Measured by Number Correct on the Digit Symbol Matching Task
Description: Change in cognitive function in the experimental group vs. controls, measured by score on the Digit Symbol Matching Task, a timed measure of attention and processing speed. Participants are asked to correctly match pairs of shapes and numbers. Scores exceeding the normative mean number correct (mean = 65.79) reflect better task performance and scores below the normative mean reflect poorer performance.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: Analysis of outcome measure excludes participants who did not complete this task / timepoint and performance-based outliers.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of correct matches
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 48 | 48
number of correct matches
  Baseline | 63.0 [61.1 to 65.0] | 63.5 [61.6 to 65.5]
  Week 6: number analyzed (Participants) | 42 | 48
  Week 6 | 67.8 [65.7 to 69.9] | 69.0 [67.0 to 70.9]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; Linear Mixed Effects Model: main effects of arm group (intervention vs. waitlist control) and timepoint (all measures from baseline to week 6), arm group x timepoint interaction. Modified intent-to-treat analysis with all participants who were randomized and completed at least the baseline study visit included in the analysis. Participants in the intervention hypothesized to improve relative to waitlist control; Test type: Superiority; p = 0.54, Mixed Models Analysis — Threshold for statistical significance: p < 0.05. Exploratory efficacy analysis - p-value not adjusted for multiple comparisons; Degrees of freedom for the group x timepoint interaction: 3, 261; Mean Difference (Final Values) = 0.12 — Linear mixed effects interaction reported for group (intervention vs. waitlist control) and timepoint (all measures baseline to week 6)

2. Secondary Outcome: Change in Daily Functioning, as Measured by the NeuroQOL Cognitive Function Scale
Description: Change in scores on the NeuroQOL Cognitive Function scale in the experimental group vs. controls. The NeuroQOL Cognitive Function scale is a 28-item self-report measure of daily functioning. Higher scores, defined as those exceeding the population mean (mean (SD) = 50.09 (10.23)), reflect better self-reported daily cognitive abilities, while lower scores, defined as those falling below the population mean, reflect poorer self-reported daily cognitive abilities.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: Analysis of outcome measure excludes participants who did not complete this scale / timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 49 | 49
score on a scale
  Baseline | 25.4 [24.3 to 26.6] | 25.7 [24.5 to 26.9]
  Week 6: number analyzed (Participants) | 44 | 48
  Week 6 | 30.2 [29.0 to 31.4] | 28.6 [27.4 to 29.8]
Statistical Analysis 1: Comparison: AKL-T01 Intervention; Linear Mixed Effects Model: main effects of arm group (intervention vs. waitlist control) and timepoint (all measures from baseline to week 6), arm group x timepoint interaction. Modified intent-to-treat analysis with all participants who were randomized and completed at least the baseline study visit included in the analysis; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 239; Mean Difference (Final Values) = 2.83 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Cognitive Performance, as Measured by Proportion Correct on the Multiple Object Tracking Test
Description: Change in scores on the Multiple Object Tracking task in the experimental group vs. controls This task measures sustained attention, cognitive control, and working memory, and requires participants to remember and track a set of target circles as they move around the screen, among a larger set of identical distractor circles. The outcome measure is the proportion of dots that a participant was able to track and identify successfully (on a scale of 0 to 1, with 0 being no dots and 1 being all of the dots). Higher proportion reflects better performance, while lower proportions reflect poorer task performance.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of dots tracked
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 47 | 49
proportion of dots tracked
  Baseline | 0.72 [0.71 to 74] | 0.73 [0.72 to 0.75]
  Week 6: number analyzed (Participants) | 44 | 49
  Week 6 | 0.78 [0.76 to 0.80] | 0.76 [0.74 to 0.78]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 229; Mean Difference (Final Values) = 0.07 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Cognitive Performance, as Measured by Digit Span on the Digit Span Backwards Test
Description: Change in scores on the Test My Brain (TMT) Digit Span Backwards task in the experimental group vs. controls. This task measures sustained attention and working memory. Participants are shown a series of numbers and asked to reproduce them in reverse order. Higher digit spans, defined as those exceeding the population mean (M = 5.98) reflect better performance, while lower digit spans reflect poorer task performance.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: digit span
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 49 | 49
digit span
  Baseline | 4.7 [4.4 to 5.1] | 4.9 [4.5 to 5.2]
  Week 6: number analyzed (Participants) | 44 | 48
  Week 6 | 5.6 [5.2 to 5.9] | 5.7 [5.3 to 6.0]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 269; Mean Difference (Final Values) = 0.89 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Cognitive Performance, as Measured by the Simple Reaction Time Test
Description: Change in scores on the Simple Reaction Time task in the experimental group vs. controls This task measures simple reaction time and psychomotor speed, and requires participants to press a key whenever a green square appears. Faster response times indicate better performance than slower response times.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millisecond
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 48 | 49
millisecond
  Baseline | 450 [431 to 470] | 434 [414 to 453]
  Week 6: number analyzed (Participants) | 44 | 48
  Week 6 | 375 [355 to 396] | 411 [392 to 431]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 236; Mean Difference (Final Values) = 5.00 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Cognitive Performance, as Measured by the Choice Reaction Time Test
Description: Change in scores on the Choice Reaction Time task in the experimental group vs. controls This task measures processing speed and cognitive control, and requires participants to indicate the direction of an arrow that is a different color from the rest. Faster response times indicate better performance than slower response times.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millisecond
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 46 | 48
millisecond
  Baseline | 1183 [1135 to 1230] | 1164 [1118 to 1211]
  Week 6: number analyzed (Participants) | 42 | 47
  Week 6 | 1062 [1013 to 1112] | 1028 [981 to 1075]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.96, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 257; Mean Difference (Final Values) = 0.11 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Cognitive Performance, as Measured by Proportion Correct on the Letter-Number Switching Test
Description: This task measures sustained attention and set-shifting, and requires participants to switch between responses to letters and numbers. The outcome measure is proportion of correct switch trials, indicating that participants successfully switched from a letter response to a number response, or vice versa (on a scale of 0 to 1, with 0 being no correct switches and 1 being correct switches on all switch trials). Higher proportion correct for switch trials indicates better set-shifting performance, while lower proportion correct indicates worse set-shifting performance.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of correct switch trials
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 47 | 48
proportion of correct switch trials
  Baseline | 0.93 [0.92 to 0.95] | 0.95 [0.94 to 0.96]
  Week 6: number analyzed (Participants) | 43 | 48
  Week 6 | 0.98 [0.96 to 0.99] | 0.96 [0.94 to 0.97]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 262; Mean Difference (Final Values) = 2.78 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change in Cognitive Performance, as Measured by D-prime on the Gradual Onset Continuous Performance Test
Description: This task measures sustained attention and response inhibition, and requires participants to respond to target stimuli and ignore distractors. Performance is measured by d-prime, a measure of memory sensitivity and discrimination. D-prime is based on the calculation of hits (i.e., responding to a target when a target is present), misses (i.e., not responding when a target is present), false alarms (i.e., responding to a target when a distractor is present), and correct rejections (i.e., not responding when a distractor is present). D-prime scores range from 0 (chance) to 4.65 (based on hit rate of 0.99 and false alarm rate of 0.01). Greater d-prime scores reflect better performance than lower d-prime scores.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: d-prime
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 48 | 49
d-prime
  Baseline | 2.3 [2.2 to 2.4] | 2.3 [2.1 to 2.4]
  Week 6: number analyzed (Participants) | 43 | 46
  Week 6 | 2.4 [2.2 to 2.5] | 2.4 [2.2 to 2.5]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.60, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 3, 227; Mean Difference (Final Values) = 0.62 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change in Cognitive Performance, as Measured by Percent Correct on the Visual Paired Associates Task
Description: Change in scores on the Visual Paired Associates Task in the experimental group vs. controls. This task measures visual memory, and requires participants to learn and identify image pairs. The outcome measure is proportion of image pairs successfully recalled (on a scale of 0 to 1, with 0 being no image pairs and 1 being all of the image pairs). A higher proportion of correct image pairs reflects better performance than a lower proportion of correct image pairs.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of image pairs
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 48 | 49
proportion of image pairs
  Baseline | 0.56 [0.52 to 0.59] | 0.56 [0.52 to 0.59]
  Week 6: number analyzed (Participants) | 44 | 48
  Week 6 | 0.60 [0.57 to 0.64] | 0.67 [0.64 to 0.70]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.06, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 1, 89; Mean Difference (Final Values) = 3.77 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Overall Daily Functioning, as Measured by the World Health Organization Disability Assessment Scale (WHODAS) 2.0
Description: Change in total score on the 36-item WHODAS in the experimental group vs. controls. The WHODAS 2.0 assesses the following domains of functioning: cognition, mobility, getting along, self-care, participation, and life activities. Scores range from 0 (no disability) to 100 (maximum disability), with higher scores reflecting a greater degree of overall functional disability.
Time Frame: Baseline and Post Treatment (6 weeks)
Population: Analysis of outcome measure excludes participants who did not complete this scale / timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AKL-T01 Intervention | Waitlist Control
Number analyzed (Participants) | 44 | 48
score on a scale
  Baseline | 70.4 [67.4 to 73.4] | 69.8 [67.0 to 72.7]
  Week 6: number analyzed (Participants) | 43 | 43
  Week 6 | 60.4 [57.3 to 63.5] | 66.1 [63.0 to 69.1]
Statistical Analysis 1: Comparison: AKL-T01 Intervention vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Degrees of freedom for the group x timepoint interaction: 1, 73; Mean Difference (Final Values) = 4.37 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected in all participants for the duration of enrollment. Adverse event data were collected for 10 weeks in: participants in the intervention arm and participants in the waitlist control arm, including control participants who did not start the intervention. Adverse event data were collected for 6 additional weeks (16 weeks total) in: control participants who started the intervention after the waitlist control arm.
Arm/Group | AKL-T01 Intervention | Waitlist Control | Control Arm Participants Who Started AKL-T01 Intervention | Control Arm Participants Who Declined AKL-T01 Intervention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/46 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/46 | 0/2
Other Adverse Events (participants affected / at risk) | 5/55 | 2/55 | 2/46 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AKL-T01 Intervention (N=55) | Waitlist Control (N=55) | Control Arm Participants Who Started AKL-T01 Intervention (N=46) | Control Arm Participants Who Declined AKL-T01 Intervention (N=2)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0) | 1 (3) | 0 (0) — Participants experienced dizziness during gameplay, particularly during fast racing sessions.
Nausea (Gastrointestinal disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) — Participant experienced nausea the seven times she played the game - reported feeling nauseous in the middle of each daily session.
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — Daily game session triggered headaches due to cognitive exertion / visual tracking.
Visual symptoms (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant had difficulty with visual sensations following gameplay.
Planned surgery (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant had planned gastrointestinal surgery during enrollment. Did not impact participation.
Fall (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant fell on ice in the park. No injury or loss of consciousness.
Cancer recurrence (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant had a recurrence of cancer during participation and opted to withdraw.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT04843930/Prot_SAP_000.pdf